CLINICAL TRIAL: NCT06855693
Title: Oral Health Care Guidance to Enhance Parent Confidence and Ability to Improve Toothbrushing Performance for Autistic Children
Brief Title: Involving Parents to Improve Tooth Brushing for Autistic Children.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sussex Community NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 331171
Record Dates: First submitted 2025-02-19; First posted 2025-03-04 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Oral Health
Keywords: oral health; children; autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Delivering better oral health: an evidence-based toolkit for prevention (Experimental): The PHE Delivering Better Oral Health toolkit has been developed with the support of the 4 UK Chief Dental Officers. This is a general population approach to Oral Hygiene advice and includes the following: Effective toothbrushing with a fluoride toothpaste is important to support oral health. The physical action of brushing removes plaque, which prevents gingivitis and periodontitis, and the fluoride in toothpaste is effective against tooth decay. The following key messages for the population include when and how to brush, specific habits associated with brushing, and, where necessary, assistance with brushing. There may be adaptations of toothbrushes, such as special grip handles, that are helpful to people who have limited manual dexterity.
  Interventions: Behavioral: Delivering better oral health: an evidence-based toolkit for prevention
- Mini Mouth Care Matters guide for special Education Settings (Experimental): Oral hygiene guidance from a Clinical standard for autistic children and young people and/or those with a learning disability in special educational settings (Mini Mouth Care Matters Special Education Settings resources. This is a specific approach to providing Oral Hygiene for children with sensory challenges. This clinical standard supports the vision of universal access whereby everyone receives quality health services that meet their specific needs. The clinical standard is designed to be used by all those involved in improving health outcomes and quality of life, including eating, speaking and socialising, for autistic children and young people, and those with a learning disability in England. It is accompanied by a supporting package of tools, resources, and modules to support the delivery of the oral healthcare assessment (either face to face or remote) and to support teams in the development o
  Interventions: Behavioral: Mini Mouth Care Matters guide for special Education Settings

INTERVENTIONS:
Behavioral: Delivering better oral health: an evidence-based toolkit for prevention — The PHE Delivering Better Oral Health toolkit has been developed with the support of the 4 UK Chief Dental Officers. This is a general population approach to Oral Hygiene advice and includes the following:
  Effective toothbrushing with a fluoride toothpaste is important to support oral health. The physical action of brushing removes plaque, which prevents gingivitis and periodontitis, and the fluoride in toothpaste is effective against tooth decay. The following key messages for the population include when and how to brush, specific habits associated with brushing, and, where necessary, assistance with brushing. There may be adaptations of toothbrushes, such as special grip handles, that are helpful to people who have limited manual dexterity.
  Arms: Delivering better oral health: an evidence-based toolkit for prevention
Behavioral: Mini Mouth Care Matters guide for special Education Settings — 2. Oral hygiene guidance from a Clinical standard for autistic children and young people and/or those with a learning disability in special educational settings (Mini Mouth Care Matters Special Education Settings resources.
  This is a specific approach to providing Oral Hygiene for children with sensory challenges.
  This clinical standard supports the vision of universal access whereby everyone receives quality health services that meet their specific needs.
  The clinical standard is designed to be used by all those involved in improving health outcomes and quality of life, including eating, speaking and socialising, for autistic children and young people, and those with a learning disability in England.
  It is accompanied by a supporting package of tools, resources, and modules to support the delivery of the oral healthcare assessment (either face to face or remote) and to support teams in the development of complementary tailored mouthcare plans.
  Arms: Mini Mouth Care Matters guide for special Education Settings

SUMMARY:
Parents of autistic children have reported a lack of understanding by oral health care staff around delivery of oral health preventive habits for their children.

This study aims to investigate if oral healthcare training utilising the Mini Mouth Care Matters (MCM) programme designed for Special Education Settings (SES) enhances parent confidence in their ability to influence their child's oral health, increases toothbrushing episodes and reduces challenging toothbrushing behaviour of autistic children.

The participants of this study will be parents of children who have a confirmed professional diagnosis of Autistic Spectrum Disorder. Parents will be recruited via healthcare professionals who provide oral health promotion within SES. Special Education Settings will be randomised into one of two groups. Group one will receive 'delivering better oral health' advice. Group two will receive the MCM user intervention guide for oral healthcare.

A maximum of 30 parents will be recruited into each intervention arm. A maximum of 60 parents will be recruited to the study.

DETAILED DESCRIPTION:
Description of the Intervention:

The first national dental health survey for special schools in England shows that:

* At ages 5 and 12, compared to previous surveys in mainstream education, the proportion of children in special education with substantial plaque visible is almost double.
* Children aged 5 in special schools were twice as likely to have had one or more teeth extracted.

The Office of the Chief Dental Officer Special Education Settings Team has developed resources which focus on prevention for better oral health for children with learning disabilities, autism or both. Resources include information and tips to help parents and carers with frequent concerns such as: Am I using the right toothpaste? Have I got the right toothbrush? Is the environment right? Am I doing it right? The resources are available on the HEE hub e- Learning for Healthcare (e-LfH) through the link Mini Mouth Care Matters (Mini MCM) Special Education Settings (SES).

The participants of this study will be parents recruited through contact with Special Educational Settings designated for oral health promotion activity from the Special Care Dental Service. Parents invited to be included in the study will be parents of children aged 3 to 15 years, with a confirmed professional diagnosis of Autistic Spectrum Disorder.

Participants will be divided by schools into two groups of parents. Each group will be randomly assigned to either the mini MCM intervention or the 'Delivering Better Oral Health' intervention. A written consent form will be provided for participants. After receiving the information regarding the study participants will be given a minimum of 48 hours to consider the information supplied before deciding whether they would like to participate. Sample size calculation based on the measure of toothbrushing performance indicates a minimum requirement of 24 participants in each group. Two groups of 30 parents will be recruited considering that children may be lost to follow-up. Group 1 parents will receive the typical model of oral health education i.e. 'Delivering Better Oral Health' intervention, providing facts about why toothbrushing should occur and advice for their child aligned with the Public Health England and Department of Health document: "Delivering better oral health: an evidence-based toolkit for prevention".

Group 2 parents will be provided with a training session using the resources developed for Mini Mouth Care Matters SES, which include specific strategies to be considered and adopted for children who are resistant to toothbrushing. The training sessions for both groups will be followed up with weekly telephone sessions for three weeks, with the option of a face-to-face visit in place of one or more telephone sessions. Both groups will receive the same Tooth Care Pack containing a selection of toothbrushes and toothpastes.

A baseline of parental attitudes using the Oral Health Behaviours Questionnaire will be recorded.

Occurrence and severity of toothbrushing behaviour problems will be recorded at baseline and at the post training intervention three week follow-up using the 13-step assessment tool identifying steps completed by parents or children, or steps not possible to complete. Parents will also be asked to record time spent toothbrushing.

Results will be analysed to examine any inter- and intra-group differences in toothbrushing behaviour and parent confidence regarding their ability to influence their child's oral health by successfully delivering twice daily toothbrushing episodes for their autistic child.

ELIGIBILITY:
Inclusion Criteria:

* Parent/Carer of an autistic child aged between 3 and 15 years Parent/Carer of an autistic child attending a Special Education Setting Parent/Carer with capacity to provide consent

Exclusion Criteria:

* Parent/Carer that cannot adequately understand verbal explanations or information written in English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
The 13-step toothbrushing assessment tool | baseline and immediately after the intervention
  The 13-step assessment tool identifies steps completed by parents or children, or steps not possible to complete. Parents will also be asked to record time spent toothbrushing.
The validated Parental-Caregiver Current Oral Health Behaviours Questionnaire (OHBQ). | baseline
  The OHBQ has been developed to measure attitudes and beliefs of parents around their child's dental health. A section to capture demographic data, with questions utilised in previous studies, has been incorporated in the questionnaire sheet above the OHBQ to explore oral health inequalities associated with socioeconomic status, which are widely observed in the literature6.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Parry, FDS RCS(Paeds) MDentSci BDS, Principal Investigator — Sussex Community NHS Foundation Trust
Locations (1):
- Sussex Community NHS Foundation Trust, Brighton, East Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: No